CLINICAL TRIAL: NCT01137227
Title: Factors Associated With Physical Inactivity Among Adolescents: a Systematic Review and Meta-analysis
Brief Title: Factors Associated With Physical Inactivity Among Adolescents
Acronym: FAPIA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Paulo Rossi Menezes, University of São Paulo, School of Medicine, Department of Preventive Medicine
Other Study IDs: FAPIA 0501/09
Record Dates: First submitted 2010-05-28; First posted 2010-06-04 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-04

CONDITIONS: Physical Inactivity; Obesity; Overweight
Keywords: Physical activity; Epidemiology; Questionnaire; Cross-sectional study
MeSH Terms: conditions — Sedentary Behavior; Obesity; Overweight; Motor Activity

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Description: 2137 studies retrieved in 8 databases (Biomed Central, CINAHL, EMBASE, ERIC, PsycInfo, PUBMED, SCOPUS, SPORTDiscus and uploaded in EndNote Web®.
  332 studies were excluded as duplicates by EndNote Web®.
  1805 titles and abstracts were assessed independently by two researchers (PG/AM): 1541 studies excluded.
  264 studies referred for full-text assessment by two independent investigators (PG/AM)
  225 studies were excluded according to the eligibility criteria (in case of discrepancies in the assessment of the researchers, studies were reviewed in duplicate)
  39 Studies assessed for quality using STROBE
  13 Studies were included in the descriptive synthesis

SUMMARY:
Despite the acknowledgment that physical activity is important for health, there are still few population-based or school-based studies that uses the current physical activity guidelines for adolescents.

Physical inactivity was defined a less than 300 min/w of moderate to vigorous-intensity physical activity practice.

Previous research has shown very high prevalence rates of physically inactive adolescents and a strong association with demographic, socioeconomic and biological factors.

Based on this information, the investigators are elaborating a systematic review of literature to obtain and provide more accurate information in this context.

DETAILED DESCRIPTION:
The objectives of this study were to (i) review extant literature on the prevalence of physical inactivity (PI) in adolescents of both sex (10-18 years old); (ii) compare its prevalence between developed and developing countries.

The search was carried out using online databases (Biomed Central, CINAHL, EMBASE, ERIC, MEDLINE, PsycInfo, Scopus, SPORTDiscus), references cited by retrieved articles and by contact with the authors, considering articles published from the establishment of the databanks until April 29th, 2010.

ELIGIBILITY:
Inclusion Criteria:

* Cross-sectional studies.
* Original studies showed that physical inactivity is evaluated through a questionnaire.
* Studies which ranked 300> inactivity min/wk.

Exclusion Criteria:

* Studies did not assess physical inactivity through a questionnaire.
* Studies in which the participants were only overweight/obese, diabetics or suffering from another disease.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Samples of adolescents (age range 10-18y) without diseases and/or physical limitations.
Sampling Method: Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Obtain the prevalence of physical inactivity in adolescents (age 10-18 y) using a questionnaire. | up than 1 week
  For the purpose of our systematic review, physical inactivity was defined as less than 300 minutes per week of moderate to vigorous physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Menezes, PhD, Principal Investigator — University of São Paulo, School of Medicine, Department of Preventive Medicine; Paulo Henrique A Guerra, Bachelor, Principal Investigator — University of São Paulo, School of Medicine, Heart Institute of General Hospital (InCor HCFMUSP), Clinical Epidemiology Unit; Augusto Cesar F de Moraes, Bachelor, Principal Investigator — University of São Paulo, School of Medicine, Children's Institute
Locations (1):
- Universidade de São Paulo, School of Medicine, São Paulo, São Paulo, Brazil